CLINICAL TRIAL: NCT05806307
Title: Comparing the Effectiveness of Misoprostol, Oxytocin, Carbetocin, Vasopressin, Bupivacaine and Epinephrine, Combined IV TXA Acid and Ethamsylate and Peri Cervical Tourniquet for the Reduction of Blood Loss During of Abdominal Myomectomy.
Brief Title: Methods Decreasing Bleeding in Open Myomectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AN2023-1
Record Dates: First submitted 2023-03-10; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Misoprostol Allergy; Oxytocin Allergy; Tranexamic Acid Allergy; Ethamsylate Allergy; Myoma; Blood Loss, Surgical
Keywords: misoprostol; oxytocin; carbetocin; tranexamic acid; ethamsylate; tourniquet; blood loss; myomectomy; vasopressin; bupivacaine; epinephrine
MeSH Terms: conditions — Myoma; Blood Loss, Surgical; Hemorrhage; Diabetes Insipidus | interventions — Misoprostol; Tourniquets; carbetocin; Oxytocin; Ethamsylate; Vasopressins; Terlipressin; Bupivacaine

STUDY DESIGN:
Intervention Model Description: Intervention
  All women will be randomly assigned to either:
  Group A (misoprostol): who will receive 800 microgram misoprostol rectally one and half hour before operation.
  Group B (Tourniquet): The operation will be performed with the use of Foleys catheter as an improvised tourniquet applied at the base of the uterus.
  Group C (Carbetocin): intramural; preparation of 100 μg of carbetocin diluted within 10 cm of saline (0.9%) Group D (Oxytocin): who will receive oxytocin 40 I.U. intramyometrially Group E (combined TXA and ethamsylate): will receive 1 g tranexamic acid and 500 mg ethamsylate IV 10 minutes before skin incision Group F receive terlipressin intramyometrial injection of one ampoule of vasopressin containing 20 units in1 ml after dilution in 19 ml of normal saline.
  Group G: infiltration of the serosa and / or myometrium with a solution composed of 50 ml Bupivacaine 0.25% and 0.5 mg of epinephrine
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- misoprostol (Active Comparator): 15 patients will receive 800 microgram (tablet 200mcg X 4) misoprostol (Misotac 200 mcg, SIGMA pharmaceutical, Egypt) rectally one and half hour before operation.
  Interventions: Drug: Misoprostol
- Tourniquet (Active Comparator): (15 patient): The operation will be performed with the use of Foleys catheter as an improvised tourniquet applied at the base of the uterus then infiltration myometrium overlying the leiomyoma with a solution composed of Bupivacaine Hcl 0.25% and 0.5 mg of epinephrine
  Interventions: Device: Tourniquet
- Carbetocin (Active Comparator): intramural; preparation of 100 μg of carbetocin ((Pabal, Ampoule 100 mcg in 1 ml, Carbetocin; FERRING, North York, Canada) diluted within 10 cm of saline (0.9%) in sterile syringe then will inject the substance into the multiple sites intramyometrial in a circumferential manner 1-2 cm away from the margins of the myoma in the planned uterine-incision site just before uterine incision for myoma extraction.
  Interventions: Drug: Carbetocin
- Oxytocin (Active Comparator): 15 patients): who will receive oxytocin 40 I.U. intramyometrially (Syntocinon, Ampule 10 I.U. in 1 ml, Oxytocin; NOVARTIS, Basel, Switzerland) then will inject the substance into the multiple sites intramyometrial in a circumferential manner 1-2 cm away from the margins of the myoma in the planned uterine-incision site just before uterine incision for myoma extraction.
  Interventions: Drug: Oxytocin
- combined TXA and ethamsylate (Active Comparator): (Patient 15): will receive 1 g tranexamic acid (2 ampoules of kapron 500 mg, kapron®, Amoun, Egypt) and 500 mg ethamsylate (2 ampoule of ethamsylate 250 mg, Dicynone, OM pharma, Geneva, Switzerland) IV 10 minutes before skin incision by slowly intravenous injection Then infusion was applied continuously for 24 hours within 1 liter of saline as 1 mg/kg/hour.
  Interventions: Drug: combined TXA and ethamsylate
- vasopressin (Active Comparator): 15 women will receive terlipressin (Glypressin, Ferring, Egypt) intramyometrial injection of one ampoule of vasopressin containing 20 units in1 ml after dilution in 19 ml of normal saline during myomectomy.
  Interventions: Drug: Vasopressin
- bupivacaine and epinephrine (Active Comparator): 15 women in which the operation will be performed after infiltration of the serosa and / or myometrium overlying the leiomyoma before uterine incision with a solution composed of 50 ml Bupivacaine Hcl 0.25% (Bucain® Weimer pharma, for Actavis Group PTC) and 0.5 mg of epinephrine Hcl (2 vials of Epinephrine® 0.25mg/1ml Misr Co. for Pharmaceutical Industries).
  Interventions: Drug: Bupivacaine Hydrochloride 0.5 % Injectable Solution epinephrine

INTERVENTIONS:
Drug: Misoprostol — (15 patient): who will receive 800 microgram (tablet 200mcg X 4) misoprostol (Misotac 200 mcg, SIGMA pharmaceutical, Egypt) rectally one and half hour before operation.
  Other Names: Misotac
  Arms: misoprostol
Device: Tourniquet — (15 patient): The operation will be performed with the use of Foleys catheter as an improvised tourniquet applied at the base of the uterus then infiltration myometrium overlying the leiomyoma with a solution composed of Bupivacaine Hcl 0.25% and 0.5 mg of epinephrine
  Other Names: Foleys catheter
  Arms: Tourniquet
Drug: Carbetocin — (15 patients): intramural; preparation of 100 μg of carbetocin ((Pabal, Ampoule 100 mcg in 1 ml, Carbetocin; FERRING, North York, Canada) diluted within 10 cm of saline (0.9%) in sterile syringe then will inject the substance into the multiple sites intramyometrial in a circumferential manner 1-2 cm away from the margins of the myoma in the planned uterine-incision site just before uterine incision for myoma extraction.
  Other Names: pabal
  Arms: Carbetocin
Drug: Oxytocin — (15 patients): who will receive oxytocin 40 I.U. intramyometrially (Syntocinon, Ampule 10 I.U. in 1 ml, Oxytocin; NOVARTIS, Basel, Switzerland) then will inject the substance into the multiple sites intramyometrial in a circumferential manner 1-2 cm away from the margins of the myoma in the planned uterine-incision site just before uterine incision for myoma extraction.
  Other Names: syntocinone
  Arms: Oxytocin
Drug: combined TXA and ethamsylate — (Patient 15): will receive 1 g tranexamic acid (2 ampoules of kapron 500 mg, kapron®, Amoun, Egypt) and 500 mg ethamsylate (2 ampoule of ethamsylate 250 mg, Dicynone, OM pharma, Geneva, Switzerland) IV 10 minutes before skin incision by slowly intravenous injection Then infusion was applied continuously for 24 hours within 1 liter of saline as 1 mg/kg/hour.
  Other Names: Kapron and Dycinone
  Arms: combined TXA and ethamsylate
Drug: Vasopressin — 15 patient intramyometrial injection of one ampoule of vasopressin containing 20 units in1 ml after dilution in 19 ml of normal saline during myomectomy.
  Other Names: Glypressin
  Arms: vasopressin
Drug: Bupivacaine Hydrochloride 0.5 % Injectable Solution epinephrine — 15 patient infiltration of the serosa and / or myometrium overlying the leiomyoma before uterine incision with a solution composed of 50 ml Bupivacaine Hcl 0.25% (Bucain® Weimer pharma, for Actavis Group PTC) and 0.5 mg of epinephrine Hcl (2 vials of Epinephrine® 0.25mg/1ml Misr Co. for Pharmaceutical Industries).
  Other Names: marcaine
  Arms: bupivacaine and epinephrine

SUMMARY:
Uterine leiomyomas (fibroids or myomas) are benign, smooth muscle tumors of the human uterus. Most myomas are asymptomatic (symptomless) and are discovered incidentally during a routine pelvic examination or imaging studies and have a lifetime incidence of approximately 70% in the general population . However, Approximately 20-40% of women with fibroids experience significant symptoms and consult gynecologic care. The most common clinical symptoms include abnormal uterine bleeding, dysmenorrhea, pelvic pain, infertility, and recurrent pregnancy loss

The standard treatment of symptomatic leiomyomas is Abdominal myomectomy Blood loss during myomectomy can be intra-operative or postoperative and with hematoma formation. The average volume of blood loss during abdominal myomectomy is 200 to 800 ml. massive blood loss associated with the dissection of huge fibroids renders myomectomy a more technically challenging procedure than hysterectomy. Sometimes myomectomy is converted to hysterectomy intra-operatively when bleeding becomes heavy and uncontrollable or when it is impossible to reconstruct the uterus because of the many defects left by removal of multiple myomas .

Many techniques are used to reduce blood loss during myomectomy; preoperative measures such as correction of preoperative anemia associated with menorrhagia may be treated with iron supplementation, use of gonadotropin (GHG) triggers prior to surgery. Intra-operative measures as use of tourniquet around the uterus during the operation, injections of Vasopressin or other vasopressors as epinephrine in the uterine muscle and use of ecbolic (misoprostol, oxytocin, and carbetocin etc.). Uterine artery ligation, embolization, or internal iliac artery ligation may also be used to avoid hysterectomy when heavy bleeding is anticipated or occurs during myomectomy

DETAILED DESCRIPTION:
The aim of study:

The aim of the study is to compare the effectiveness of a single preoperative dose of rectal misoprostol, intramyometrial oxytocin, intramyometrial carbetocin, combined iv TXA acid and ethamsylate and peri cervical tourniquet for the reduction of blood loss during of abdominal myomectomy.

Methodology:

Type of Study: Prospective randomized comparative clinical trial Study Setting: This study will be conducted in Cairo University, kasr al-ainy hospitals, Maternity hospital in operative theater.

Study Period: 6 months from April 2023 to October 2023. Study Population: Patients will be recruited in this study from those attending gynecology ward at Kasr al-ainy hospitals, Maternity hospital who are 25-48 years old with symptomatic uterine myoma indicating operative management, abnormal uterine bleeding or bulk-related symptoms, females with infertility or recurrent pregnancy loss, pressure symptoms, and large myoma(s).

Basic assessment:

* Verbal consent was obtained before history taking All women were subjected to
* Detailed clinical history.
* Personal history:

Name, Age, Parity, Occupation, Residency and Special habits.

· Present history: History of onset, course and duration of agonizing symptoms, history of HMB, history of infertility, history of pelvic pain.

• Obstetric history: History of previous abortion, ectopic pregnancy, previous cesarean section and interval between cesarean deliveries.

· Menstrual history: Age of menarche and LMP.

· Past history: History of medical disorders, drug therapy or allergy, history of appendicitis - in particular, appendix rupture, history of exposure to radiation treatment for cancer, history of Gynecological infections (PID), history of abdominal infections e.g.: peritonitis, history of any abdominal or pelvic operation for non-obstetric cause.

• Family history: Family history of uterine myoma, family history of uterine cancers. Examination

* General examination includes blood pressure, heart rate, body temperature, head& neck examination, chest, heart, sign of anemia, height (in cm) and weight (in kg) measurements to calculate the Body mass index (The formula for BMI is weight in kilograms divided by height in meters squared).
* Local clinical examination: assessment of maternal health, abdominal and bimanual examination, speculum examination to roll out any vaginal or cervical infection and local cause of bleeding.
* Preoperative investigations (Complete blood picture, blood group, RH, Kidney Function Test , Liver Function Test , random Blood Sugar , urine analysis, Coagulation profile).
* Ultrasonography examination (abdominal / vaginal) and MRI: to assess the following data:

Presence of uterine myoma, size and site of myoma, uterine size, roll out any adnexal mass.

Intervention

All women will be randomly assigned to either:

Group A (misoprostol) (25 patient): who will receive 800 microgram (tablet 200mcg X 4) misoprostol (Misotac 200 mcg, SIGMA pharmaceutical, Egypt) rectally one and half hour before operation.

Group B (Tourniquet) (25 patient): The operation will be performed with the use of Foleys catheter as an improvised tourniquet applied at the base of the uterus close to the insertion of the uterosacral ligaments a minor hole through the broad ligament on either side of the uterus will be made, the catheter will be passed through the two holes and knotted firmly anteriorly around the uterus, the tourniquet will be tensed in stepwise manner by alternatively holding with a clamp, pulling on the tourniquet, and again holding with another clamp in such a way that it temporarily impedes the blood supply from the uterine vessels. The fallopian tubes, the ovaries, and the infundibulopelvic ligament are kept away to avoid compression by tourniquet then operation will be performed after infiltration of the serosa and / or myometrium overlying the leiomyoma before uterine incision with a solution composed of 50 ml Bupivacaine Hcl 0.25% (Bucain® Weimer pharma, for Actavis Group PTC) and 0.5 mg of epinephrine Hcl (2 vials of Epinephrine® 0.25mg/1ml Misr Co. for Pharmaceutical Industries). The solution will be prepared just before the procedure. Before each infiltration, aspiration will be performed to avoid intravascular injection.

Group C (Carbetocin) (25 patients): intramural; preparation of 100 μg of carbetocin ((Pabal, Ampoule 100 mcg in 1 ml, Carbetocin; FERRING, North York, Canada) diluted within 10 cm of saline (0.9%) in sterile syringe then will inject the substance into the multiple sites intramyometrial in a circumferential manner 1-2 cm away from the margins of the myoma in the planned uterine-incision site just before uterine incision for myoma extraction.

Group D (Oxytocin) (25 patients): who will receive oxytocin 40 I.U. intramyometrially (Syntocinon, Ampule 10 I.U. in 1 ml, Oxytocin; NOVARTIS, Basel, Switzerland) then will inject the substance into the multiple sites intramyometrial in a circumferential manner 1-2 cm away from the margins of the myoma in the planned uterine-incision site just before uterine incision for myoma extraction.

Group E (combined TXA and ethamsylate) (Patient 25): will receive 1 g tranexamic acid (2 ampoules of kapron 500 mg, kapron®, Amoun, Egypt) and 500 mg ethamsylate (2 ampoule of ethamsylate 250 mg, Dicynone, OM pharma, Geneva, Switzerland) IV 10 minutes before skin incision by slowly intravenous injection Then infusion was applied continuously for 24 hours within 1 liter of saline as 1 mg/kg/hour.

The operations will be performed by the same team to avoid any bias related to surgical skills. The abdomen will be exposed through Pfannenstiel incision, after skin incision, the subcutaneous fat and abdominal fascia will be opened crosswise, and the rectus muscle will be opened on the midline. The parietal peritoneum will be opened longitudinally to reach the pelvic cavity. Subsequently, a self-retaining retractor will be inserted, and intestine will be packed. Uterus will be inspected for the number, location, and shape of myomas, and other pelvic organs will be inspected for associated pathology. Uterine incisions on top of myoma will be performed. When possible, uterine incisions will be performed on the anterior wall or the fundus in order to reduce postoperative adhesions. The incision will be performed using monopolar diathermy. Intracapsular enucleation of myomas will be performed by gently dissecting between the myoma and the pseudo capsule. The myoma will be grasped by Collins forceps and gently enucleated out. Meticulous hemostasis will be secured by low-voltage coagulation (≤30 W) of feeding vessels. Myoma bed will be closed by 1 or 2 layers (The uterine defects will be closed with sutures in layers. If the myometrial defect is deep (>2 cm), two layers may be needed to approximate the tissue and achieve hemostasis) of interrupted vicryl sutures (Vicryl 1-0 polyglactin 910; Egycryl, Taisier CO, Egypt). The serosa is closed with a running suture; we used size 2-0 polyglactin 910 (Vicryl). At the end of the surgery, 1 intraperitoneal suction drain will be routinely used and the volume in the drain bag will be measured every 12 hours. (Ultramed, Nelaton drain-24 FG, Assiut City, Egypt). in all patients the drains will be removed on the second postoperative day unless otherwise indicated. Number and size of myomas will be recorded. Myoma size represent the mean size of each myoma. Enucleated myomas will be sent to histopathology.

Total bleeding was calculated as intraoperative and postoperative blood loss. Intraoperative blood loss was estimated by the scrub nurse by drying up all blood in the surgical field with swabs and then weighing them. The weight of the dry surgical swabs (roughly 28 g for each 30 * 30 cm abdominal swabs) is measured before use and after being wet or soaked by blood. A highly accurate digital balance is used to measure the weight in grams. The weight difference is translated into the blood loss considering that 1 g is equal to 1 mL blood. The quantity of blood loss (mL) equals (weight of the used materials - weight of the materials prior to the surgery) in addition to the blood collected in the suction apparatus after evacuation. Meanwhile, postoperative blood loss was defined as the blood volume found in the suction drain.

All study groups will be checked for vital signs (blood pressure, heart rate, and respiratory rate) before and after myomectomy. The following routine investigations, CBC, PT, PTT, ALT, AST and serum creatinine, will be performed preoperatively for all groups, and CBC will be repeated on the third postoperative day. Any adverse effects in either group will be recorded. The need for blood transfusion either intraoperatively or postoperatively will be also recorded. Intraoperative blood transfusion will be governed by clinical condition and amount of blood loss. Postoperative blood transfusion will be indicated if hemoglobin (Hb) percentage was less than 7 g/dl with relevant clinical manifestations. Women will be reviewed again 1 week after the operation. In addition to the usual follow-up, women will be checked for manifestations of thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged between 25 to 48 years old.
2. BMI less than 35 kg/m2
3. symptomatic uterine myomas..
4. myoma staging from (3 to 6) according to FIGO staging through trans vaginal ultrasonography (TVUSG) or magnetic resonance imaging (MRI) according to FIGO classification.
5. Maximum diameter of the largest myoma is 15 cm.
6. Uterine size between 14 to 28 weeks pregnancy.

Exclusion Criteria:

1. History of previous myomectomy
2. Allergy to Misoprostol, carbetocin, TXA, ethamsylate, Oxytocin, vasopressin, bupivacaine and epinephrine.
3. Hypertension.
4. Cardiac and Pulmonary diseases.
5. Patients who have bleeding disorders.
6. Patients on antiplatelets or anticoagulant before surgery.
7. Anemia (Hb < 10g %).
8. Chronic endocrine or metabolic diseases such as Diabetes.
9. Renal and hepatic impairment.
10. Obesity (body mass index > 30 kg/m2).
11. Cases that will require intraoperative conversion of myomectomy to hysterectomy.
12. Intracavitary, submucosal, pedunculated Subserosal and adnexal Myoma FIGO staging 0,1,2,7,8.
13. history of Gynecological infections (PID), history of abdominal infections e.g.: peritonitis, history of any abdominal or pelvic operation for non-obstetric cause.

Ages: 25 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients will be recruited in this study from those attending gynecology ward at Kasr al-ainy hospitals, Maternity hospital who are 25-48 years old with symptomatic uterine myoma indicating operative management, abnormal uterine bleeding or bulk-related symptoms, females with infertility or recurrent pregnancy loss, pressure symptoms, and large myoma(s).
Enrollment: 105 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
blood loss | 3 hours
  the estimated intra-operative blood loss in ml

SECONDARY OUTCOMES:
blood transfusion | 24 hours
  Number of patients in each group who require transfusion and how many units they need
Preoperative and postoperative hemoglobin values | 48 hours
  will be measured in g/dl on 24 hours before and 24 hours after surgery
Perioperative blood pressure | 4-6 hours
  Measure blood presure in mmhg at start and end of operation and then every hour interval up to first four hours postoperative
the duration of hospital stays | 3 day
  How many days patient stay in hospital after surgery for recovery
Operation time | 3 hours
  measured from incision of first myoma to serosal closure of last myoma wound in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Taymour, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine, Kasr el ainy hospital, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper JM, Brady RM. Intraoperative and early postoperative complications of operative hysteroscopy. Obstet Gynecol Clin North Am. 2000 Jun;27(2):347-66. doi: 10.1016/s0889-8545(00)80026-1. PMID 10857125
- [Background] Donnez J, Dolmans MM. Uterine fibroid management: from the present to the future. Hum Reprod Update. 2016 Nov;22(6):665-686. doi: 10.1093/humupd/dmw023. Epub 2016 Jul 27. PMID 27466209
- [Background] Kongnyuy EJ, Wiysonge CS. Interventions to reduce haemorrhage during myomectomy for fibroids. Cochrane Database Syst Rev. 2014 Aug 15;2014(8):CD005355. doi: 10.1002/14651858.CD005355.pub5. PMID 25125317
- [Background] Krentel H, De Wilde RL. Complications in Laparoscopic Supracervical Hysterectomy(LASH), especially the morcellation related. Best Pract Res Clin Obstet Gynaecol. 2016 Aug;35:44-50. doi: 10.1016/j.bpobgyn.2015.11.001. Epub 2015 Nov 14. PMID 26694587
- [Background] Mohamed, S. E. S., Mansour, D. Y., & Shaker, A. N. (2019). The effect of misoprostol on intra-operative blood loss during myomectomy operation: Randomized controlled trial. Evidence Based Women's Health Journal, 9(1), 363-371.
- [Background] Shady, N. W., Sallam, H. F., & Fahmy, H. (2018). Reducing blood loss during open myomectomy with intravenous versus topical tranexamic acid: A double-blinded randomized placebo-controlled trial. Middle East Fertility Society Journal, 23(3), 225-231.
- [Background] Sirkeci RF, Belli AM, Manyonda IT. Treating symptomatic uterine fibroids with myomectomy: current practice and views of UK consultants. Gynecol Surg. 2017;14(1):11. doi: 10.1186/s10397-017-1014-4. Epub 2017 Jul 6. PMID 28890674
- [Background] Sleiman Z, Baba RE, Garzon S, Khazaka A. The Significant Risk Factors of Intra-Operative Hemorrhage during Laparoscopic Myomectomy: A Systematic Review. Gynecol Minim Invasive Ther. 2019 Nov 11;9(1):6-12. doi: 10.4103/GMIT.GMIT_21_19. eCollection 2020 Jan-Mar. PMID 32090006
- [Background] M Al-Morsi, A., N Abdul-Galeel, K., & A El-Desouky, E. S. (2021). Comparative study between oxytocin versus tranexamic acid and ethamsylate combination in reducing intraoperative blood loss in myomectomy. Al-Azhar Medical Journal, 50(3), 1893-1908.
- [Result] Camanni M, Bonino L, Delpiano EM, Ferrero B, Migliaretti G, Deltetto F. Hysteroscopic management of large symptomatic submucous uterine myomas. J Minim Invasive Gynecol. 2010 Jan-Feb;17(1):59-65. doi: 10.1016/j.jmig.2009.10.013. PMID 20129334